CLINICAL TRIAL: NCT06781905
Title: Description of Neurocognitive and Psychiatric Disorders Associated With Targeted Therapies Used in the Treatment of Lung Cancers With ALK/ROS1 Fusion and Their Impact on Patients' Quality of Life: Construction of an Experimental Patient-researcher Collaborative Care and Research Pathway
Acronym: DRACONIS
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0158; 2024-A02274-43 (Other: ID-RCB)
Record Dates: First submitted 2025-01-08; First posted 2025-01-17 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Lung Cancer; Metastatic Lung Cancer With ALK/ROS1 Fusion
Keywords: Neurocognitive disorders; Targeted therapies; Quality of life; Lung cancer; Collaborative research; Care pathway
MeSH Terms: conditions — Lung Neoplasms; Neurocognitive Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with ALK/ROS1-positive lung cancer treated with anti-ITK-ALK/ROS1 reporting neurocognitive: Patients presenting a cognitive and/or neuropsychiatric complaint (i.e. patients reporting a subjective loss of their cognitive abilities and/or the appearance of neuropsychiatric symptoms) and/or patients identified by a carer or relative as presenting cognitive impairment and/or neuropsychiatric symptoms.
  Interventions: Other: Assessments of neuropsychiatric, neurocognitive and psychosocial alterations

INTERVENTIONS:
Other: Assessments of neuropsychiatric, neurocognitive and psychosocial alterations — Assessments will be conducted over two consecutive days or on a separate visit, depending on participant preferences and logistical constraints. The first day will focus on the evaluation of neuropsychiatric and neurocognitive alterations. A comprehensive assessment involving various tools will be carried out by a psychiatrist, a neuropsychologist, and a neurologist. The second day, which may take place on-site or remotely (by telephone or secure videoconference), will be dedicated to psychosocial assessments by a team of social psychologists using a comprehensive qualitative and quantitative approach to quality of life: daily life management, social relationships, and self-image and self-esteem. The collected data will be subjected to a reflexive thematic analysis. The qualitative exploration of quality of life will be complemented by a quantitative assessment using a standardized tool (EORTC QLQ LC13 and C30).

SUMMARY:
Targeted cancer therapies have a higher therapeutic index than chemotherapy and are prescribed to tens of thousands of patients in France each year. These treatments modify often ubiquitous signaling pathways involved in neuronal synaptic plasticity, the cellular substrate of cognitive and psychiatric functions. Neurocognitive and psychiatric disorders associated with targeted therapies are poorly described and therefore still poorly understood, although they appear to be clinically more severe than chemobrain (neurocognitive disorders related to chemotherapy).

The case of patients with metastatic lung cancer with ALK/ROS1 fusion is emblematic. These cancers are treated very effectively with oral targeted therapies inhibiting the tyrosine kinase activity of ALK or ROS1 proteins (ITK-ALK/ROS1), with survival that can exceed 10 years. However, neurocognitive and psychiatric disorders associated with anti-ITK-ALK/ROS1 are reported in 7 to 60% of patients, with a prevalence of about 10% with anti-ITK-ALK/ROS1 brigatinib or alectinib and up to 53% with lorlatinib in industrial therapeutic trials. These disorders appear to be particularly frequent and severe with lorlatinib, including cognitive disorders - especially memory - mood disorders such as anxiety, depression and emotional lability, and psychotic disorders. Current therapeutic trials and care pathways are not designed to take into account these side effects related to anti-ITK-ALK/ROS1. Their incidence is therefore probably underestimated.

The DRACONIS project aims to:

(1) describe the complaints +/- neurocognitive and neuropsychiatric disorders associated with anti-ITK-ALK/ROS1 through a rigorous neuropsychological and psychiatric evaluation (i.e. patient phenotyping) and (2) understand the experience of complaints +/- neurocognitive and neuropsychiatric disorders associated with anti-ITK-ALK/ROS1 and their consequences on patients' quality of life in a comprehensive approach.

The DRACONIS project is part of a multidisciplinary and collaborative approach through the establishment of a partnership between researchers, clinicians and representatives of the anti-ITK-ALK/ROS1 France Cancer du Poumon patient association. The project is notably monitored by a joint scientific committee composed of researchers, clinicians, patients and patient caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older, fluent in French
* Currently treated with anti-ITK-ALK/ROS1 for ALK/ROS1-positive lung cancer
* Identified by the prescribing physician as having complaints with or without associated neurocognitive and/or neuropsychiatric disorders related to the treatment.

Exclusion Criteria:

* History of neurocognitive and/or neuropsychiatric disorders prior to initiation of anti-ITK-ALK/ROS1 targeted therapy, excluding disorders associated with anti-ITK-ALK/ROS1 or other systemic anticancer treatments
* Patients with uncontrolled brain metastases or carcinomatous meningitis (requiring symptomatic treatment with corticosteroids progressive or symptomatic)
* Patients who do not have sufficient proficiency in French to complete questionnaires and/or participate in semi-structured interviews
* Severe, progressive or unstable medical conditions that may interfere with the evaluation variables (uncontrolled epilepsy, acute psychiatric or psychotic disorders, visual hallucinations, acute infection).
* Consumption of toxic substances that may affect cognitive performance
* Deafness or blindness that may compromise participant evaluation or participation in tasks and scales
* Patients who refuse to participate in the study or are unable to express thein non-opposition to participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ALK/ROS1-positive lung cancer treated with anti-ITK-ALK/ROS1
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2027-05-09 (Estimated); Study Completion 2027-05-09 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive and neuropsychiatric characterization of patients on anti-ITK-ALK/ROS1 targeted therapy who reported treatment-releated neurocognitive and/or neuropsychiatric complaints or disorders | From enrollmenet day 1 visite to the end of the participation, day 2.
  Exploratory and comprehensive approach to neurocognitive and neuropsychiatric disorders that may be experienced by patients treated with anti-ALK/ROS1 targeted therapy for ALK/RO1 lung cancer. The characterization of complaints with or without associated neurocognitive and/or neuropsychiatric disorders will be achieved by combining the results of neuropsychological assessments and psychiatric evaluations.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Day care Hospital, Pierre Wertheimer Hospital, Civil Hospitals of Lyon, Bron
  - Pneumology service, Louis Pradel Hospital, Civil Hospitals of Lyon, Bron

IPD SHARING:
Plan to Share IPD: Undecided